CLINICAL TRIAL: NCT02326636
Title: Fecal Microbiota Transplant for Recurrent Clostridium Difficile Infection
Acronym: FMT
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Nimisha Parekh, Associate Clinical Professor, University of California, Irvine
Other Study IDs: 20139455
Record Dates: First submitted 2014-12-09; First posted 2014-12-29 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A donor stool sample will be kept for future testing in case of contamination.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Fecal Microbial Transplantation — Participants with refractory Clostridium difficile infection will be given healthy donor stool administered by colonoscopy or enema.

SUMMARY:
The purpose of this research is to investigate the efficacy of transplanting screened donor fecal material in treating patients with recurrent Clostridium difficile infection. Participants with refractory Clostridium difficile infection will be given healthy donor stool administered by colonoscopy or enema and their response will be evaluated by symptom questionnaire and stool testing for Clostridium difficile at 4 weeks after the treatment.

ELIGIBILITY:
Inclusion Criteria for Recipient:

* Between the age of 18 and 100
* Have positive Clostridium difficile polymerase chain reaction (PCR) or toxin
* Have symptoms of > 3 watery loose stools a day for at least 2 consecutive days
* Have failed at least one prior standard course of antibiotic therapy.

Examples of standard therapy are:

* Metronidazole 500 mg three times a day for 10 to 14 days
* Vancomycin 125 mg four times a day for 10 to 14 days
* Not be pregnant and have negative urine and/or serum human chorionic gonadotropin (hCG) test
* Not be taking oral or intravenous steroids in the past three months.
* Not on biologic agents, anti-tumor necrosis factor (anti-TNF) agents, cyclosporine, mercaptopurine, azathioprine, methotrexate or chemotherapy in the preceding 3 months
* Not have profound immunosuppression: Chemotherapy the preceding 3 months, HIV/AIDS, decompensated cirrhosis
* Not be in the Intensive Care Unit
* Not be a transplant recipient

Exclusion Criteria for Recipient:

* Not between the age of 18 and 100
* Does not have positive Clostridium difficile PCR or toxin
* Does not have symptoms of > 3 watery loose stools a day for at least 2 consecutive days
* Has not failed at least one prior standard course of antibiotic therapy. Examples of standard therapy are:
* Metronidazole 500 mg three times a day for 10 to 14 days
* Vancomycin 125 mg four times a day for 10 to 14 days
* Is pregnant
* Has taken oral or IV steroids in the past three months.
* Has taken biologic agents, anti-TNF agents, cyclosporine, mercaptopurine, azathioprine, methotrexate or chemotherapy in the preceding 3 months
* Has profound immunosuppression: Chemotherapy the preceding 3 months, HIV/AIDS, decompensated cirrhosis
* In the Intensive Care Unit
* Is a transplant recipient

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are referred for recurrent Clostridium difficile infections. Donors will be identified by the Recipient.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2014-04; Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
The recurrence rate of Clostridium difficile 4 weeks after FMT. | Four weeks

SECONDARY OUTCOMES:
Clinical symptoms from before fecal microbiota transplant (FMT) to 4 weeks after FMT. | Four weeks
Satisfaction with the FMT procedure. ( satisfaction questionnaire ) | Up to 24 weeks
  Subjects will complete a satisfaction questionnaire following the FMT procedure.
Quality of life before and 4 weeks after FMT. | Four weeks
  Subjects will complete a quality of life questionnaire before and 4 weeks after FMT.
Alternate treatments needed for Clostridium difficile before and after FMT. | Up to 24 weeks
  Subjects medication and treatment history for Clostridium difficile before and after FMT will be collected.
The rate of adverse events that may be related to FMT. | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nimisha Parekh, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States